CLINICAL TRIAL: NCT02949687
Title: Duodenal Ileal Interposition With Sleeve Gastrectomy and Selective Intra-Abdominal Denervation for Type 2 Diabetes Mellitus
Brief Title: Surgical Treatment in Diabetic Patients With Grade 1 Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator institution change
Sponsor: Universidade Positivo (Other)
Responsible Party: Principal Investigator, Luciana El-Kadre, invited clinical professor, Universidade Positivo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 37048114.9.0000.0093
Record Dates: First submitted 2016-10-21; First posted 2016-10-31 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus; Obesity
Keywords: ileal interposition; metabolic surgery; diabetes; intra abdominal selective denervation
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Sympathectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ileal interposition sleeve sympathectomy (Experimental): laparoscopic ileal interposition with sleeve and sympathectomy
  Interventions: Procedure: ileal interposition with sleeve and sympathectomy

INTERVENTIONS:
Procedure: ileal interposition with sleeve and sympathectomy — laparoscopic ileal interposition with sleeve and sympathectomy

SUMMARY:
Surgical Treatment in Diabetic Patients With Grade 1 Obesity

DETAILED DESCRIPTION:
There will be a randomized clinical trial, non-blind, 1-arm treatment (Duodenal Ileal Interposition with Sleeve Gastrectomy and Selective Intra-Abdominal Denervation for Type 2 Diabetes Mellitus), including 40 research subjects with type 2 diabetes mellitus and obesity class I. In order to analise the effect on weight loss and glycemic control after 2 years of follow up

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of type 2 diabetes mellitus
* Both sexes were treated with oral antidiabetic agents and / or insulin except the current treatment with Glucagon-like peptide-1 (GLP-1) receptor agonists or dipeptidyl peptidase 4 inhibitors
* Stable antidiabetic medication within the last 8 weeks prior to randomization (V2), if therapy includes insulin, the average daily dose should not have changed by more than 10% in the past 8 weeks
* HbA1c> 8.0%
* Age> 20 years and <60 years
* Body mass index (BMI) of 30 35 kg / m²
* Agree to sign the consent form

Exclusion Criteria:

* Type 1 diabetes mellitus (positive for anti-GAD), or GAD negative anti anti body with low β cell function (C-peptide after stimulation <0.5 ng / ml)
* Current treatment with GLP-1 receptor agonist and / or dipeptidyl peptidase 4 inhibitors
* Recent vascular event (myocardial infarction, coronary angioplasty or stroke in the past 6 months)
* Malignant neoplasm
* Portal hypertension
* Inability to cooperate with segment
* Low capacity of understanding surgery
* Unrealistic expectations of the outcome
* Cognitive impairment
* Current pregnancy
* Moderate or severe mood disorder; severe anxiety; eating disorders (based on Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria)
* Chemical dependency or alcoholism (based on DSM-V criteria).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
glycated hemoglobin(HbA1c) level of 6.0% or less, without the use of diabetes medications | 2 YEARS
  Success Rate of Biochemical Resolution of Diabetes at 24 Months as Measured by HbA1c ≤ 6% With no Diabetes Medications

IPD SHARING:
Plan to Share IPD: No